CLINICAL TRIAL: NCT02434263
Title: A Clinical Evaluation of the HYDRA Self Expanding Transcatheter Aortic Valve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vascular Innovations Co. Ltd. (Industry)
Collaborators: MedPass International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VI-CL-HYDRA-02
Record Dates: First submitted 2015-04-27; First posted 2015-05-05 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydra TAVI (Experimental): Percutaneous Replacement of the Diseased Aortic Valve
  Interventions: Device: Hydra TAVI

INTERVENTIONS:
Device: Hydra TAVI — Percutaneous Replacement of the Diseased Aortic Valve
  Other Names: TAVR

SUMMARY:
The purpose of this study is the evaluation of the performance, safety and efficacy of Hydra Aortic valve in real-world patients. Following initial implantation, all patients will have clinical follow up at 30 days, 3, months, 6 months and 12 months

DETAILED DESCRIPTION:
This study is a multicenter, prospective, non-randomized investigational study designed to assess the safety and performance of the HYDRA Aortic valve and delivery system. Primary endpoint for safety is the 30 day all cause mortality rate. Primary endpoint for performance is the acute device success. In addition, the efficacy of the HYDRA Aortic valve and delivery system will be evaluated. Up to 165 patients will be enrolled in the study in order to achieve 150 subjects successfully implanted.

All patients will have a clinical follow-up at 30 days, 3months, 6 months and 12 months post implant. The follow-up procedure table is shown in Appendix A.

The patient is enrolled in the study as a subject only upon signature of the informed consent. All subjects will be reviewed by the Principal Investigator prior to undergoing the implant procedure for the Hydra Aortic Heart Valve.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has given written Informed Consent for study participation prior to procedure.
2. Greater than 55 years of age.
3. Aortic annulus diameter meets the range 18 to 27mm as measured by CT conducted within the past 180 days, or echocardiogram (TEE 3D recommended) if medically contraindicated to CT.
4. Patient has severe degenerative aortic stenosis with echocardiography derived mean gradient >40mmHg and/or peak velocity greater than 4.0 m/s and/or an initial valve area of <1.0 cm2.
5. Patient has symptomatic aortic stenosis as demonstrated by NYHA Functional Classification of II or greater.
6. Patient is deemed high operable risk and suitable for TAVI.
7. Patient's predicted operative mortality or serious, irreversible morbidity risk is <50% at 30 days.
8. Patient has structurally normal cardiac anatomy.
9. Willing and able to comply with all required follow-up evaluation

Exclusion Criteria:

1. Patient has a history of a cerebral vascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months.
2. Patient has carotid artery disease requiring intervention.
3. Patient has evidence of a myocardial infarction (MI) within the past 6 months.
4. Patient has hypertrophic cardiomyopathy.
5. Patient has a native aortic valve that is congenitally uni-cuspid, bicuspid, quadricuspid or non-calcified as seen by echocardiography.
6. Patient has mitral or tricuspid valvular regurgitation (≥ grade III) or moderate to severe mitral stenosis.
7. Patient has aortic root angulation >70 degrees (horizontal aorta).
8. Patient has aortic root diameter of < 26 mm or >36 mm.
9. Patient has a pre-existing prosthetic valve or prosthetic ring in any position.
10. Patient refuses blood transfusion or surgical valve replacement.
11. Patient has resting left ventricular ejection fraction (LVEF) < 20%.
12. Patient has documented, untreated symptomatic coronary artery disease (CAD) requiring revascularization.
13. Patient has severe basal septal hypertrophy.
14. Patient has had a percutaneous interventional or other invasive cardiac or peripheral procedure ≤ 14 days of the index procedure (does not apply for diagnostic angiography or Angio-CT).
15. Patient has a history of or has active endocarditis.
16. Patient has echocardiographic evidence of intracardiac mass, thrombus, or vegetation.
17. Patient has hemodynamic instability (requiring inotropic support or mechanical heart assistance).
18. Patient is in acute pulmonary edema or requiring intravenous diuretic therapy to stabilize heart failure.
19. Patient with significant pulmonary disease (FEV1 < 30% as predicted).
20. Patient has significant chronic steroid use as determined and documented by the Principal Investigator.
21. Patient has a known hypersensitivity or contraindication to anticoagulant or antiplatelet medication.
22. Patient has renal insufficiency as evidenced by a serum creatinine > 3.0 mg/dL (265.5μmol/L) or end-stage renal disease requiring chronic dialysis.
23. Patient's iliofemoral arteries have severe calcification, tortuosity (>two 90 degree bends), diameter <6mm, or subject has had an aorto-femoral bypass that preclude safe placement of a 18 French sheath.
24. Patient has blood dyscrasia (leukopenia, acute anemia, thrombocytopenia, bleeding diathesis, or coagulopathy).
25. Patient has a current autoimmune disease that, in the opinion of the Principal Investigator precludes the subject from study participation.
26. Patient has significant aortic disease.
27. Patient has a pre-existing endovascular stent graft in the supra- or infrarenal aorta or pre-existing stent grafts in the iliofemoral arteries.
28. Patient has an active peptic ulcer or has had gastrointestinal (GI) bleeding within the past 90 days prior to procedure
29. Patient has a life expectancy < 12 months.
30. Patient has other medical, social or psychological conditions that, in the opinion of the Principal Investigator, preclude the subject from study participation.
31. Patient has a known allergy to contrast media, nitinol alloys or bovine tissue.
32. Patient has a history of any cognitive or mental health status that would interfere with study participation.
33. Currently participating in another trial.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2015-08-13 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 30 days
  30-day mortality of procedure is defined as all deaths occurred in subjects attending the Hydra prosthesis implantation within 30 days post procedure. All deaths include in-hospital mortality, cardiac death, valve-related death, and death of unknown cause

SECONDARY OUTCOMES:
Procedural Success | 3, 6, and 12 months
  Composite outcome measures consisting of Effective orifice area, mean aortic valve gradient, degree of prosthetic valve regurgitation.

CONTACTS AND LOCATIONS:
Locations (6):
- General Hospital of Athens Ippokration, Athens, Greece
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Vilnius University Hospital Santariškiu Klinikos, Vilnius, Lithuania
- Waikato Hospital, Hamilton, New Zealand
- Instytut Kardiologii im.Prymasa, Warsaw, Poland
- King Chulalongkorn Hospital, Bangkok, Thailand

REFERENCES:
- [Derived] Aidietis A, Srimahachota S, Dabrowski M, Bilkis V, Buddhari W, Cheung GSH, Nair RK, Mussayev AA, Mattummal S, Chandra P, Mahajan AU, Chmielak Z, Govindan SC, Jose J, Hiremath MS, Chandra S, Shetty R, Mohanan S, John JF, Mehrotra S, Sondergaard L. 30-Day and 1-Year Outcomes With HYDRA Self-Expanding Transcatheter Aortic Valve: The Hydra CE Study. JACC Cardiovasc Interv. 2022 Jan 10;15(1):93-104. doi: 10.1016/j.jcin.2021.09.004. PMID 34991828